CLINICAL TRIAL: NCT01694017
Title: Economic Evaluation of Treatment of HIV With Zidovudine/Stavudine and Tenofovir Regimen: A Cost Effectiveness Study
Brief Title: Economic, Clinical and Quality of Life Assessment in Patients on Antiretroviral Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Christian Medical College, Vellore, India (Other)
Responsible Party: Principal Investigator, Christine A. Wanke, Professor of Medicine and Public Health and Community Medicine, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10465
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: HIV
Keywords: HIV,treatment,cost effectiveness,drug toxicity,QOL,costs
MeSH Terms: interventions — Tenofovir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zidovudine (Active Comparator): zidovudine 300 mg + lamivudine 150 mg + nevirapine 200 mg , once daily, for a year
  Interventions: Drug: Zidovudine
- Tenofovir (Active Comparator): tenofovir 300 mg+ emtricitabine 200 mg + efavirenz 600 mg, once daily, for one year
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — tenofovir 300 mg+ emtricitabine 200 mg + efavirenz 600 mg, once daily, for one year
  Other Names: Atripla; Vonavir
  Arms: Tenofovir
Drug: Zidovudine — zidovudine 300 mg + lamivudine 150 mg + nevirapine 200 mg , once daily, for a year
  Other Names: Lazid-N; Duovir-N; Zidolam-N
  Arms: Zidovudine

SUMMARY:
The purpose of this study is to compare clinical, economical and quality of life (QOL) outcomes in patients living with HIV on zidovudine/stavudine regimen and tenofovir regimen. This study will be an unblinded randomized trial. The first step will be empirical data collection for one year for calculating the incremental cost effectiveness ratio (ICER). The second step will be to perform a simulation model for calculating long term ICER.

DETAILED DESCRIPTION:
The drug regimen for treatment of HIV at the free ART centers in India includes stavudine/zidovudine and lamivudine with nevirapine. Approximately 20-30% of the patients on this regimen experience drug toxicity within the first six months of treatment.

The tenofovir based regimen is one of the least toxic regimens with less than 5% of patients experiencing toxicity. Tenofovir based regimen is not considered as the first choice for ART in the Indian governmental program, because it is more expensive than the other drug regimens, in spite of better clinical outcomes in resource limited settings. The cost of treatment with stavudine/zidovudine is presumed to be less expensive and is the preferred first line treatment, but we believe that although the direct cost to the government is less, patients on zidovudine/stavudine regimen have to spend more money for additional hospital visits and admissions, laboratory investigations and other medications due to ART induced toxicity.

There are no published data including economic, clinical and quality of life outcomes to compare the two regimens from India. Hence, this unblinded randomized pragmatic comparative effectiveness study will seek to identify the best treatment for HIV patients based on the incremental cost effectiveness ratio (ICER), quality of life (QOL) and clinical outcomes.

The clinical outcomes include viral suppression, change in the CD4 and proportion of patients with toxicity and opportunistic infections. Direct costs for the treatment will be calculated. The QOL scores will be estimated and compared between the regimens using questionnaires. QOL scores and direct cost will be used as utilities for calculating ICER.

ELIGIBILITY:
Inclusion Criteria:

* All treatment naïve patients above 18 years confirmed with the diagnosis of HIV
* Eligible for initiation of cART based on the National Aids Control Organization of India
* Consenting for participation and follow-up for one year.

Exclusion Criteria:

* All patients requiring hospitalization at the time of initiation of treatment
* Patients with opportunistic infections including tuberculosis
* Patients with co-morbidities like diabetes or neurological impairments
* Pregnant and breast feeding women and children less than 18 years will be excluded
* All patients living outside the catchment area of CMC and not willing for regular follow-up will be excluded
* Patients with a creatinine clearance less than 50 mL/min will be excluded.
* Patients receiving other co-medications with possible interaction with tenofovir, like antifungal (voriconazole), ergot derivatives (dihydroergotamine, ergonovine, ergotamine, and methylergonovine), benzodiazepines (midazolam, triazolam), calcium channel blocker (bepridil), GI motility agent (cisapride), neuroleptic (pimozide) and St.John's wort will be excluded.
* Patients with hemoglobin less than 8 gm/dl
* Patients started on tenofovir regimen by the treating physician at the time of enrollment will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Viral suppression | End of follow-up : end of 12th Month
Change in CD4 levels | End of Months 6 and 12
Drug related toxicity | Months : 1,2,3,4,5,6,7,8,9,10,11,12
opportunistic infections | Months: 1,2,3,4,5,6,7,8,9,10,11,12
Direct costs | Months: 1,2,3,4,5,6,7,8,9,10,11,12
Quality of life | Month 1 and end of months 4,8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Wanke, MD, Study Chair — Tufts University; Sowmyanarayanan V Thuppal, MD, Principal Investigator — Tufts University
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India